CLINICAL TRIAL: NCT07083050
Title: Connective Tissue Graft vs Volume Stable Collagen Matrix (Geistlich Fibro-Gide®) for Coverage of Multiple Gingival Recession Defects in Combination With Coronally Advanced Flap (CAF) Randomized Multicenter Controlled Clinical Trial Assessing Non-Inferiority in Root Coverage
Brief Title: Non-Inferiority of Fibroguide Collagen Membrane Compared to Autologous Connective Tissue Graft for Coverage of Multiple Adjacent Recession. Multicenter Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maurizio Tonetti (Network)
Collaborators: University of Florence (Other); Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor-Investigator, Maurizio Tonetti, Executive Director, The European Research Group on Periodontology (ERGOPerio)
Organization: The European Research Group on Periodontology (ERGOPerio) (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fibroguide
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gingival Recession, Plastic Surgery
Keywords: Gingival recession; Root coverage; Collagen Construct; Connective tissue graft; Morbidity
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coronally Advanced Flap plus Collagen Matrix (Experimental): Coronally Advanced Flap plus Collagen Matrix Tissue Substitute
  Interventions: Device: Volume stable collagen matrix
- Coronally Advanced Flap plus Autologous Connective Tissue Graft (Active Comparator): Current standard of care
  Interventions: Procedure: Autologous Connective Tissue Graft from the Hard Palate

INTERVENTIONS:
Device: Volume stable collagen matrix — Volume stable collagen matrix obtained from porcine collagen after proprietary cross-linking by device manufacturer
  Other Names: Fibrogide
  Arms: Coronally Advanced Flap plus Collagen Matrix
Procedure: Autologous Connective Tissue Graft from the Hard Palate — Autologous connective tissue surgically harvested from the hard palate and transplanted in the area of gingival recession
  Other Names: CTG
  Arms: Coronally Advanced Flap plus Autologous Connective Tissue Graft

SUMMARY:
This study deals with coverage of multiple denuded roots. The current standard treatment requires surgical correction and uses soft tissue taken from the roof of the mouth to enhance results. The hypothesis of this trial is that a synthetic collagen matrix (called Fibrogide) can be used to replace soft tissue taken from the subject. If the collagen matrix will prove to be equally as effective as the patient own tissue, it will be possible to avoid a more extensive surgery and decrease pain and discomfort.

DETAILED DESCRIPTION:
Objectives Primary objective: to assess non-inferiority of differences in root coverage of recession defects comparing the use of Volume Stable Collagen Matrix (VCMX, Geistlich Fibro-Gide®) ed to the use of CTG at 12 months Secondary objectives: to assess if VCMX is non-inferior in terms of complete root coverage, percentage of root coverage and professional evaluation of aesthetics. Moreover, the study is also designed to test if VCMX Geistlich Fibro-Gide® reduces morbidity, shortens time to recovery and improves patient based related outcomes with respect to the use of autologous connective tissue graft harvested from the patient own palate when used to obtain root coverage of multiple adjacent gingival recessions. Moreover, as adverse events, complete root coverage, and professional evaluation of aesthetics will be assessed

Design and Outcomes This will be a parallel group, controlled, assessor-blind, randomized, multicenter, multinational, clinical trial.

The statistical design will be a non-inferiority trial in terms of the professional outcomes measuring root coverage and aesthetics and a superiority trial in terms of patients related outcomes.

Based on a recently completed and published RCT with similar design (Geistlich Mucograft® study), the sample size has been estimated in 80 subjects per treatment arm (about 200 recessions/arm) to be analyzed with a multilevel statistical approach and a non-inferiority margin of 0.25 mm in recession coverage. The non-inferiority margin has been set as 50% of the clinically relevant difference estimated at 0.5 mm.

Randomization will be performed by computer generated random codes, using random permuted blocks with a block size of 4 to avoid uneven splits and minimization for the key prognostic factor cigarette smoking. Allocation will be concealed to the surgeons until completion of preparation of the recipient bed by opaque envelopes. A central study registrar will perform patient registration.

Study locations will include academic centers and a practice-based research network in Italy, Germany, and Spain.

A single examiner, blind with respect to the treatment assignment, will perform all primary outcome measurements at each center. Trained personnel not involved with the surgical intervention will: i) administer patient questionnaires, ii) provide instructions and collect patient diaries. A single calibrated investigator with specific experience in using the specific score will centrally perform assessment of esthetic scores on standardized digital images.

A biostatistician blind with respect to treatment assignment will perform the analysis.

Interventions and Duration The two intervention groups will consist of surgery with connective tissue graft from the palate (standard of care control) and surgery with the application of Geistlich Fibro-Gide®. Experienced clinicians will deliver treatment consisting of root coverage surgery using coronally advanced flaps, the most utilized procedure for coverage of multiple recessions. Surgery will be standardized and the same procedures/materials will be employed to ensure consistency essentially as performed in the completed Mucograft study.

The total duration of the Followfollow-up of individual patients will be up to 1 year and extended to 3 years for the collection of long-term follow-up data.

Sample Size and Study Population Study population will consist of 160 subjects with a minimum of two adjacent RT1 and RT2 (with periodontal attachment <2 mm) recessions of the gingival margin (average 2.5 recessions per subject, of which one should be 3 mm or deeper) requiring surgical intervention for root coverage. Heavy smokers (>10 cigarette/day) will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18 to 70 years of age, with a minimum of two adjacent teeth with gingival recession (at least one with a depth ≥ 3 mm - RT1 or RT2 with 2 mm or less of interdental periodontal attachment loss) in anterior and premolar teeth in the maxilla and requiring surgical intervention, without medical contraindications to elective surgery. In case of recessions on five or more adjacent teeth, the teeth at the external sides will not be included in the study.
* At least 2 mm marginal keratinized tissue width and irrespective of soft tissue thickness prior therapy. The study should involve treatment naïve patients in terms of root coverage procedures. Prior therapy should include treatment of gingival inflammation, if present, instructions in non-traumatic oral hygiene, and reconstruction of the cemento-enamel junction with adhesive dental materials in case of cervical abrasion or erosion involving this structure
* Evidence of subject ability to achieve good oral hygiene and control gingivitis in the whole of the dentition (FMPS<25% and FMBS<25%)
* Ability to understand study procedures and to comply with them for the entire length of the study. Ability and willingness to give written informed consent.

Exclusion Criteria:

* Presence of untreated periodontitis
* Persistence of uncorrected gingival trauma from tooth brushing
* Interdental attachment loss greater than 2 mm or furcation involvement in the experimental teeth
* Presence of less than 2 mm of keratinized tissue width
* Presence of severe tooth malposition, rotation or clinically significant super-eruption
* Self reported current smoking exceeding 10 cigarettes/day or pipe or cigar smoking
* Rheumatoid arthritis or known sensitization to collagen based medical products.
* Presence of medical contraindications to elective surgery
* Participation in another interventional clinical trial
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual to give written informed consent.
* Uncontrolled diabetes mellitus
* Allergy to collagen
* Pregnancy or lactation or sexually active female subjects who are of childbearing potential and who are not using hormonal or barrier methods of birth control (e.g., oral or parenteral contraceptives, diaphragm plus spermicide, condoms).
* Radiotherapy
* immunosuppressive therapy
* chronic steroid therapy (inhaler or systemic).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Root coverage | 12 months
  Difference in reduction in gingival recession (root coverage) between baseline and 12 months

SECONDARY OUTCOMES:
Complete root coverage | 12 months
  Frequency of teeth and subjects with complete coverage of exposed root surface
Time to recovery | The first two post-operative weeks
  Time necessary for remission of post-surgical pain and discomfort
Oral Health Related Quality of Life | 3, 6, 12, 24, and 36 months
  Oral Health Impact Profile (OHIP-14) instrument - Scale 0-10 with higher scores indicating a better outcome

OTHER OUTCOMES:
Tissue thickness | 6 and 12 months
  Marginal soft tissue thickness measured digitally on intraoral scan

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD PhD, Principal Investigator — The European Research Group on Periodontology (ERGOPerio)
Locations (2):
- Ospedale Careggi, Florence, Italy
- International University of Catalunya, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided